CLINICAL TRIAL: NCT05174130
Title: Evaluation of the Therapeutic Usability of RESPIRA ADVANCED Device in Patients Under Invasive Mechanical Ventilation in Stable Phase and in Weaning Phase
Brief Title: Evaluation of the Therapeutic Usability of RESPIRA ADVANCED Device in Patients Under Invasive Mechanical Ventilation
Acronym: RESPIRA-02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESPIRA-02
Record Dates: First submitted 2021-11-08; First posted 2021-12-30 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: 15 patients in stable phase and 15 patients in weaning phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing mechanical ventilation in stable phase (Experimental): 15 Patients will be changed from a basal reference ventilator to the RESPIRA ADVANCED device. The patient will be ventilated for the next 24 hours with the investigational medical device or until one withdrawal criteria is met according to clinical investigation plan. After 24 hours of ventilation with the investigational medical device, the patient will be changed to the previous conventional ventilation device.
  Interventions: Device: RESPIRA device.com® Advanced
- Patients undergoing mechanical ventilation in weaning phase (Experimental): 15 Patients will be changed from a basal reference ventilator to the RESPIRA ADVANCED device. The patient will be ventilated for the next 24 hours with the investigational medical device or until one withdrawal criteria is met according to clinical investigation plan. After 24 hours of ventilation with the investigational medical device, the patient will be changed to the previous conventional ventilation device.
  Interventions: Device: RESPIRA device.com® Advanced

INTERVENTIONS:
Device: RESPIRA device.com® Advanced — Ventilation of patients with continuous monitoring of the patient's clinical parameters and the parameters that the investigational medical device shows.

SUMMARY:
The objective of the clinical investigation presented is to guarantee the safety and usability of the RESPIRA ADVANCED medical device in patients undergoing mechanical ventilation in the ICU, both stable patients and in the weaning phase. Through the clinical investigation, the reliability and durability of the device, the adequacy of the ventilatory parameters and their consistency over time, and the response of the patients wills be checked. During the entire course of the patient's participation in the study, the patient will be closely monitored following the protocol specifications, to guarantee safety and evaluate the effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Availability of a family member or legal representative capable of understanding and signing the informed consent
* Patient admitted to the intensive care unit requiring invasive mechanical ventilation, who shows:
* Hemodynamic stability: MAP ≥ 65 mmHg and norepinephrine requirements ≤ 0.5 µg / kg / min, and
* Respiratory stability: PaO2 / Fraction of Inspired Oxygen (FiO2)> 100 and stable oxygen requirements in the previous 6 hours.
* In case is considered to start phase of "weaning" or awakening, the level of sedation should allow adequate triggering of the inspiratory trigger, in a patient with improvement of respiratory failure and / or radiological image.

Exclusion Criteria:

* Age under 18 years
* Weight less than 50 kg
* Body weight greater than 120 kg
* Height greater than 1,90 m
* Presence of barotrauma (pneumothorax) or pleural fistula
* Hemodynamic instability (MAP < 65 mmHg or norepinephrine requirements > 0,5 µg /kg / min)
* Neurocritical patient
* Obstetric patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate blood oxygen pressure (PaO2) changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes in PaO2 during the ventilation of the patient

SECONDARY OUTCOMES:
Evaluate the failure of the device | This variable will be analyzed at the end of the study (36 hours)
  Amount of patients that required the use of the conventional ventilator due to a therapeutic failure of the investigational device
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 0.33 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 0.66 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 2 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 4 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 8 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 12 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 16 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 20 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the tidal volume of the device | This variable will be measured and recorded at 24 hours
  Evolution of the tidal volume during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 0.33 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 0.66 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 2 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 4 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 8 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 12 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 16 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 20 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the peak pressure of the device | This variable will be measured and recorded at 24 hours
  Evolution of the peak pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 0.33 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 0.66 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 2 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 4 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 8 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 12 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 16 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 20 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the plateau pressure of the device | This variable will be measured and recorded at 24 hours
  Evolution of the plateau pressure during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 0.33 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 0.66 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 2 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 4 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 8 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 12 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 16 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 20 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the breathing rate of the device | This variable will be measured and recorded at 24 hours
  Evolution of the breathing rate during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the inspiration-expiration ratio of the device in the weaning patient's arm | This variable will be measured and recorded at 8 hours
  Evolution of the inspiration-expiration ratio during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the inspiration-expiration ratio of the device in the weaning patient's arm | This variable will be measured and recorded at 16 hours
  Evolution of the inspiration-expiration ratio during the ventilation of the patient in hours
Evaluate the reliability and temporal consistency of the inspiration-expiration ratio of the device in the weaning patient's arm | This variable will be measured and recorded at 24 hours
  Evolution of the inspiration-expiration ratio during the ventilation of the patient in hours
Evaluate the pH changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes of pH during the ventilation of the patient
Evaluate the blood carbon dioxide pressure (PaCO2) changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes of PaCO2 during the ventilation of the patient
Evaluate the oxygen saturation changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes of oxygen saturation during the ventilation of the patient
Evaluate the heart rate changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes of heart rate during the ventilation of the patient
Evaluate the breathing rate changes of patients during the ventilation procedure compared to baseline ventilation | This variable will be analyzed at the end of the study (36 hours)
  Significant changes of breathing during the ventilation of the patient
Safety Assessment | This variable will be analyzed at the end of the study (36 hours)
  Number of device related serious and unexpected adverse events reported during the use of the device
Protective Measures Assessment | This variable will be analyzed at the end of the study (36 hours)
  Number of alarms activated by the investigational device during the ventilation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Josep María Nicolás Arfelis, Principal Investigator — Hospital Clinic of Barcelona
Locations (3):
- Spain (3):
  - Hospital Universitari Germans Trias y Pujol, Badalona, Barcelona
  - Clínica Nostra Senyora del Remei, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No